CLINICAL TRIAL: NCT05594160
Title: Process Factors in Inpatient Psychotherapy
Brief Title: Agentic Self-view as Common Factor in Psychotherapy - Self-efficacy in the Treatment of Inpatients Over the Course of Time
Acronym: AGENTIC
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Simone Jennissen, Dr. phil. M. Sc., University Hospital Heidelberg
Other Study IDs: Agency-Inpatient-2022
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Inpatient Psychotherapy; Self Efficacy; Group Cohesion; Treatment Outcome
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Psychotherapy — Patients treated at the inpatient psychotherapy unit of a University Hospital receive 8 to 10 weeks of multimodal psychotherapeutic treatment. Treatment consists of individual as well as group psychodynamic therapy. Additionally, patients receive an individual combination of music, art, relaxation and body-oriented group therapy. Therapeutic treatment is provided by a multiprofessional, interdisciplinary team of psychotherapists with either a medical or psychology degree, art and music therapists, specialist nurses, social workers and physiotherapists.

SUMMARY:
The purpose of this study is to assess the development of self-efficacy over the course of psychotherapeutic inpatient treatment and to examine the interplay of symptom severity with group cohesion and positive self-view, respectively. Moreover, variables that potentially moderate the relationship between positive self-view and treatment outcome will be investigated.

DETAILED DESCRIPTION:
In this study, the aim is to investigate the role of patients' self-efficacy in inpatient psychotherapeutic treatment. More specifically, it will be explored whether patients' positive self-view over the course of psychotherapeutic treatment is linked to symptom severity throughout and at the end of inpatient treatment. Moreover, the interplay between positive self-view and other variables that could potentially influence the psychotherapeutic process such as patients' group cohesion will be investigated. Therefore, it will be examined whether changes in positive self-view and in group cohesion precede and explain symptom change. Furthermore, another objective of the study is to examine whether certain patient characteristics influence the relation between positive self-view and treatment outcome. More precisely, it will be investigated whether patient characteristics such as attachment style and tendency to self-criticism act as potential moderator variables. It is expected that positive self-view as well as stronger group cohesion will lead to subsequent symptom improvement. Additionally, it is expected that reciprocal relations between symptom severity with both positive self-view and group cohesion will be found.

For the above described purposes, data of ca. 1500 adult patients will be used that has been obtained over the course of an (usually) 8-week inpatient psychotherapeutic treatment in the years 2015 to 2021 in Heidelberg University Hospital. Patients filled in pre- as well as post-treatment questionnaires of psychotherapy outcome measures and took part in weekly questionnaire assessments of clinically relevant process variables over the course of treatment. Therefore, data analysis will be performed using the described longitudinal panel data.

To examine the influence of positive self-view on symptom severity as well as the interplay of self-view and group cohesion random-intercept cross-lagged dynamic panel models (RI-CLPM) will be used. To investigate potential moderator variables of the relation between self-efficacy and treatment outcome moderated multilevel regression models will be calculated.

Thus, the general aim of this study is to shed more light on process variables and patient characteristics that might play a role in the psychotherapeutic inpatient treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients of at least 18 years of age
* included in inpatient psychotherapy treatment program in a hospital for psychosomatic medicine
* provided measurements of symptoms, self-view, and group cohesion for at least one measurement occasion

Exclusion Criteria:

* bipolar, acute psychotic or substance abuse disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients being treated at the inpatient unit of University Hospital Heidelberg, department for psychosomatic medicine.
Sampling Method: Non-Probability Sample
Enrollment: 1544 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Symptom Checklist Short Form (SCL-K11) | Weekly assessment of each patient over the course of an (usually) 8-week inpatient psychotherapy treatment program. Data will be reported for 6 years of continuous study enrolment.
  Symptom measure assessing depressive and anxiety related symptoms with 11 items

SECONDARY OUTCOMES:
Inpatient and day clinic experiences questionnaire (IDES) - Subscale Positive Self | Weekly assessment of each patient over the course of an (usually) 8-week inpatient psychotherapy treatment program. Data will be reported for 6 years of continuous study enrolment.
  Subscale assessing patients' sense of themselves by measuring self-efficacy and self-evaluation
Inpatient and day clinic experiences questionnaire (IDES) - Subscale Group Cohesion | Weekly assessment of each patient over the course of an (usually) 8-week inpatient psychotherapy treatment program. Data will be reported for 6 years of continuous study enrolment.
  Subscale assessing the quality of the relationships between patients in an inpatient psychotherapy program

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Dinger-Ehrenthal, Prof. Dr., Study Director — Department of Psychosomatic Medicine and Psychotherapy, Medical Faculty, Heinrich-Heine University Düsseldorf

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because study data is provided by mental health patients and is therefore subject to strict protection.